CLINICAL TRIAL: NCT07089810
Title: Digital Intervention Based on BCW Theory Has a High Blood Pressure in High-risk Population of Stroke Study on the Effect of Stress on Self-management Behavior of Patients
Brief Title: Effect of Digital Intervention on Self-management of Hypertensive Patients at High Risk of Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025-K116-01
Record Dates: First submitted 2025-07-22; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-06

CONDITIONS: Hypertension; Mhealth
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital intervention has a high blood pressure in the high-risk population of stroke Study (Experimental): The chronic disease management App developed by the Affiliated Hospital of Nantong University was used to digitally manage hypertension patients, construct personalized intervention programs for such patients, and implement effective supervision and management on the platform. By strengthening the cognition of the population on the disease, it can increase their ability to self-management health, promote the change of health behavior, and ultimately reduce the incidence of stroke
  Interventions: Device: Digital intervention has a high blood pressure in the high-risk population of stroke Study on the effect of stress on self-management behavior of patients
- The control group was given health education according to the community management routine of the 20 (No Intervention): Patients in the control group will receive routine hypertension management in the community according to the recommendations of the Chinese Guidelines for the Prevention and Treatment of Hypertension (2024), including health education, lifestyle intervention, blood pressure monitoring, and regular follow-up **, but without the use of digital chronic disease management App.

INTERVENTIONS:
Device: Digital intervention has a high blood pressure in the high-risk population of stroke Study on the effect of stress on self-management behavior of patients — Intervention group (n = 60) : Interventions were developed for five behavioral problems, as follows:
  1. Lack of knowledge about hypertension
     - Measures: APP push knowledge (risk factors, medication, lifestyle, etc.), blood pressure monitoring teaching, monthly online lectures, regular feedback and encouragement of blood pressure data.
  2. Poor medication compliance
     - Measures: Medication reminders were set by the APP, and repeated and recorded when no medication was taken.
  3. Obesity/overweight Targets: BMI 18.5-23.9, waist circumference <90cm in men and <85cm in women Interventions: promoting knowledge about the dangers of obesity, daily exercise reminders, setting weight loss goals and encouraging weight loss.
  4. A high-sodium diet Target: <6g salt per day
     - Measures: Release of low-salt dietary guidelines (graphic and text) and distribution of salt-limiting spoons (1-2 grams).
  5. Drinking too much Target: ≤25g alcohol per day for men and ≤15g for women; Weekly male ≤140g, female ≤80
  Arms: Digital intervention has a high blood pressure in the high-risk population of stroke Study

SUMMARY:
Stroke is the second leading cause of death in the world, and the number of stroke patients in China ranks the first in the world. Hypertension is the most important risk factor. Studies have shown that 80% of stroke can be prevented by controlling risk factors. However, the management level of hypertension patients in China is still low, and their self-management ability is insufficient.

Digital health management, such as remote monitoring, AI and mobile health platforms, provides a new way for hypertension prevention and control. Foreign studies have shown that digital interventions can effectively improve patients' self-management behaviors, such as diet, exercise and blood pressure control. Interventions based on wechat, APP and other tools in China have also achieved positive results, but face challenges such as patient acceptance, system adaptation and data continuity.

Based on behavior change wheel (BCW) theory ** and digital platform, this study formulated personalized intervention programs for hypertension patients in high-risk groups of stroke, and promoted health behavior change from three aspects of ** ability, motivation and opportunity **. By improving disease cognition and strengthening self-management, the incidence of stroke can be ultimately reduced, and a new strategy for hypertension prevention and control in the community can be provided.

ELIGIBILITY:
Inclusion criteria:

(1) hypertensive patients at high risk of stroke screened in the National Screening and Intervention Project for High-risk Population of Stroke (2) willing to participate Cooperate and sign the informed consent form

Exclusion criteria:

(1) TIA and stroke patients (2) severe cognitive impairment (MMSE≤9) and (3) inability to use smartphones (4) Refusal to participate

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Hypertension Self-Management Behavior Rating Scale (HPSMBRS) | From the beginning of enrollment to the end 6 months later
Hypertension Knowledge Scale (HK-LS) | From the beginning of enrollment to the end 6 months later
Stroke premonitory symptom alertness assessment questionnaire | From the beginning of enrollment to the end 6 months later
Self-rating Depression Scale (PHQ-9) | From the beginning of enrollment to the end 6 months later
Generalized Anxiety Disorder-7 (GAD-7) | From the beginning of enrollment to the end 6 months later

SECONDARY OUTCOMES:
Blood Pressure (mmHg) | From the beginning of enrollment to the end 6 months later
Blood lipid (mmol/L) | From the beginning of enrollment to the end 6 months later
Fasting blood glucose (mmol/L) | From the beginning of enrollment to the end 6 months later
Glycosylated hemoglobin (HbA1c)(%) | From the beginning of enrollment to the end 6 months later
Blood homocysteine (Hcy) (mmol/L) | From the beginning of enrollment to the end 6 months later
Is the risk of stroke reduced? : Risk prediction for atherosclerotic cardiovascular disease in China Prediction for ASCVD Risk in China, China-PAR | From the beginning of enrollment to the end 6 months later

IPD SHARING:
Plan to Share IPD: No